CLINICAL TRIAL: NCT06958523
Title: Apple Health Study
Status: Recruiting | Type: Observational
Sponsor: Apple Inc. (Industry)
Collaborators: Brigham and Women's Hospital (Other); MCRA (Industry)
Responsible Party: Principal Investigator, Calum A. MacRae, Vice Chair for Scientific Innovation, Department of Medicine, Brigham and Women's Hospital
Other Study IDs: Pro00081895; 2024P003608 (Other: Brigham and Women's Hospital IRB)
Record Dates: First submitted 2025-03-05; First posted 2025-05-06 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Mental Health; Sleep; Exercise; Hormones; Metabolic Health; Hearing; Aging; Lifestyle Factors; Functional Capacity; Neurological Conditions; General Health; Wellbeing; Women's Health
Keywords: Apple Health Study; Large Scale Digital Study; Digital Biomarkers; Research App; Apple Research App; iPhone
MeSH Terms: conditions — Psychological Well-Being; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Apple Health Study aims to build a diverse and inclusive group of participants to help researchers advance our understanding of how signals and information collected from apps and devices relate to health and may be used to predict, detect, monitor, and manage changes in health.

To enroll, US residents who have an iPhone can download the Apple Research app from the App Store and go through the introduction and informed consent for the Apple Health Study. This study is fully remote, and all are invited to enroll if the eligibility criteria are met.

Participants will be asked to complete tasks and surveys, using their iPhone and Apple Research app which include:

* Selecting the types of data they would like to share with the study such as health and sensor data
* Completing tasks and surveys including areas such as personal demographic information, personal medical history, family history, and social determinants of health

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old (at least 19 years old in Alabama and Nebraska, at least 21 years old in Puerto Rico);
* Live in the United States of America;
* Have an iPhone;
* Have installed Apple Research app on your iPhone;
* Be comfortable communicating in written and spoken English;
* Be willing and able to provide informed consent to participate in the Study.

Exclusion Criteria:

* Share your iCloud account, iPhone, or devices that collect health data such as Apple Watch with anyone else, because it could result in sharing another person's health information with the Study, making it challenging for researchers to use your information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Study aims to enroll a large and representative group of at least 500,000 participants across the United States of America willing to contribute information about health and wellness over time.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Health Status | Baseline and every 6 months until study end (up to 5 years)
  Assessed by participant self-report as well as clinical health records and claims data. The initial count and change over time in the number and type of health conditions such as cardiovascular, circulatory, cognition, hearing, mental health, metabolic, mobility, neurologic, respiratory, sex and gender, reproduction, hormones, sleep, and health events such as hospitalizations, procedures or falls.

SECONDARY OUTCOMES:
Participant Population: Demographic Characteristics of Study Participants | Baseline and annually until study end (up to 5 years)
  Results of surveys to report participant demographics.
Social Determinants of Health: Lifestyle & Environment Survey | Baseline and every 6 months until study end (up to 5 years)
  Results of surveys that collect information about social determinants of health.
Family Health History in Health Conditions and Health Events | Baseline and have option to update if needed (up to 5 years)
  Results of self-reported family health history of first-degree biologic family.

CONTACTS AND LOCATIONS:
Overall Officials: Calum MacRae, MD, PhD, Principal Investigator — Brigham and Women's Hospital; Tiffany Avery, MD, Principal Investigator — MCRA
Locations (2):
- United States (2):
  - MCRA, Washington D.C., District of Columbia
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- See also: Apple Health Study Website — https://applehealthstudy.bwh.harvard.edu/